CLINICAL TRIAL: NCT06985433
Title: Light Treatment of Symptomatic Vulvovaginitis
Brief Title: Light Treatment of Vaginal Infections in Reproductive Age Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UVISA Health ApS (Industry)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uvisa03.01
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Bacterial Vaginosis; Vulvovaginal Candidiases
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment of BV with single session of light treatment. (Experimental): A group of 10 patients will receive light therapy in single treatment session to evaluate its safety and efficacy.
  Interventions: Device: Vaginal light therapy - Once
- Treatment of BV with two sessions of light treatment. (Experimental): A group of 10 patients will receive light therapy in two treatment sessions to evaluate its safety and efficacy.
  Interventions: Device: Vaginal Light Therapy - Twice
- Treatment of VVC with single session of light treatment. (Experimental): A group of 10 patients will receive light therapy in single treatment session to evaluate its safety and efficacy.
  Interventions: Device: Vaginal Light Therapy - Once
- Treatment of VVC with two sessions of light treatment. (Experimental): A group of 10 patients will receive light therapy in two treatment sessions to evaluate its safety and efficacy.
  Interventions: Device: Vaginal Light Therapy - Twice

INTERVENTIONS:
Device: Vaginal light therapy - Once — Vaginal light therapy device will deliver UVA and blue light to target symptom causing microbes in single treatment session.
  Arms: Treatment of BV with single session of light treatment.
Device: Vaginal Light Therapy - Once — Vaginal light therapy device will deliver UVA and blue light to target symptom causing microbes in single treatment session.
  Arms: Treatment of VVC with single session of light treatment.
Device: Vaginal Light Therapy - Twice — Vaginal light therapy device will deliver UVA and blue light to target symptom causing microbes in two treatment sessions.
  Arms: Treatment of BV with two sessions of light treatment.
Device: Vaginal Light Therapy - Twice — Vaginal light therapy device will deliver UVA and blue light to target symptom causing microbes in two treatment sessions.
  Arms: Treatment of VVC with two sessions of light treatment.

SUMMARY:
Antimicrobials have helped in managing vaginal dysbiotic conditions such as bacterial vaginosis (BV) and vulvovaginal candidiasis (VVC). However, their increasing inefficiency and rise in antimicrobial resistance (AMR) is a challenge and threat to public health. Therefore, this study will investigate the safety and efficacy of light as an antimicrobial to treat vulvovaginal infections.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) and vulvovaginal candidiasis (VVC) are two of the most common vaginal infections, affecting millions of women worldwide. These infections can cause significant discomfort, reduced quality of life, and, in some cases, negative reproductive outcomes. Despite their prevalence, challenges remain in accurate diagnosis, effective treatment, and long-term management, highlighting the need for new treatment methods and solid clinical evidence. BV occurs when there is an imbalance in the normal vaginal microbiota with symptoms of vaginal discharge and irritation. BV also increases the risk of sexually transmitted infections and negative pregnancy outcomes. Treatments with antibiotics have varying effectiveness and high recurrence rates. VVC is caused by an overgrowth of Candida albicans and presents as itching, burning, and thick, cottage cheese-like discharge. Although antifungal medications are often effective, recurrent VVC (RVVC) is a significant challenge requiring long-term treatment. There is also a risk of resistance to antibiotic and antifungal medications.

Self-diagnosis and self-treatment are common, which can lead to misdiagnosis and ineffective treatment. Overuse of antimicrobial medications can cause side effects and resistance. Therefore, there is a need for new treatment methods to improve patient outcomes and quality of life. This clinical trial represents a first in human pilot, efficacy study of the effectiveness of vaginal light therapy in women with BV and/or VVC. The study will also evaluate the safety and tolerability of the treatment, as well as examine the underlying vaginal microbial dynamics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years of age
* Normal gynecological status
* Diagnosed for BV or VVC
* Not pregnant
* No signs of other genital tract infections

Exclusion Criteria:

* Current signs of other genital tract infection including STD
* Concomitant medication for treatment of vaginal infections or use of any intravaginal medication during the clinical investigation
* Pregnancy
* Current genital malignancies, chemotherapy for any reason within the last 6 months, previous radiotherapy in the genitourinary system. Cervical dysplasia diagnosis or treatment within the last 3 months (where applicable)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Patient reported reduction in symptoms of BV/VVC | Upto 2 months
  Patient-reported symptoms of BV and VVC will be recorded before and after the treatment through a vaginal health questionnaire to evaluate the efficacy of light treatment based on the following scale:
  Symptom severity: 0 - 4, Lower the score, better the outcome Impact on everyday life: 0 - 4, Lower the score, better the outcome

SECONDARY OUTCOMES:
Clinical resolution of BV and/or VVC | Upto 2 months
  Patients will be examined for the objective signs of BV and VVC post treatment.
Healthier vaginal microbiome as compared to pre-treatment state. | Upto 2 months
  Vaginal swabs will be collected to evaluate vaginal microbiome dynamics before and after the treatment.
Vaginal health questionnaire | 2 Weeks
  User experience of the device will be evaluated using the vaginal health questionnaire and following scale:
  Device Use Experience: 0 - 4, Lower the score, better the outcome

OTHER OUTCOMES:
No visual sign of tissue damage from light treatment. | Upto 2 months
  Safety of the light treatment will be evaluated by visual evaluation of vulva and vagina at post treatment follow ups.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified data related to primary and secondary outcomes, which are aggregated in tabular or graphical form.
Access Criteria: Qualified researchers presenting a proposal for data use and approved scientific/clinical study plan can request access by contacting the Sponsor. Data sharing is subject to data use agreement to protect participant's confidentiality and the sponsor's proprietary interests.